CLINICAL TRIAL: NCT02834052
Title: A Phase I/II Trial of Pembrolizumab (MK-3475) and Poly-ICLC in Patients With Metastatic Mismatch Repair-proficient (MRP) Colon Cancer
Brief Title: Pembrolizumab + Poly-ICLC in MRP Colon Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Asha Nayak (Other)
Collaborators: Oncovir, Inc. (Industry); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor-Investigator, Asha Nayak, Director, Inpatient Oncology Service, Augusta University
Organization: Augusta University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCC-16047
Record Dates: First submitted 2016-06-15; First posted 2016-07-15 (Estimated); Results first posted 2024-06-07 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: Metastatic Colon Cancer; Solid Tumor
Keywords: Immunotherapy; Anti-programmed death 1 (PD-1) inhibitor; Immunostimulant; monoclonal antibody; TLR3 agonist; Immunologic factors
MeSH Terms: conditions — Colonic Neoplasms; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab; poly ICLC

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase 1 (Experimental): This "Run In" phase is aimed to determine if poly-ICLC can be safely combined with standard dosages of pembrolizumab:
  i. Pembrolizumab will be administered 200 mg intravenously (IV) every 3 weeks (q3w)
  ii. Poly-ICLC will be administered intramuscularly (IM) twice weekly at one of two dose levels: 1 mg or 2 mg
  Each dose level will enroll 3-6 participants, up to 12 participants total, depending on the occurrence of dose limiting toxicities (DLT) at each dosing level.
  Participants may receive treatment for 1 year (~17 cycles).
  Interventions: Drug: pembrolizumab; Drug: Poly-ICLC
- Phase 2 (Experimental): In Phase 2, all participants will receive the standard pembrolizumab dose (200 mg IV q3w) in addition to the maximum tolerated dose of poly-ICLC (either 1 mg or 2 mg), as determined by the Phase 1 arm.
  Up to 30 participants will be treated in Phase 2. Participants may receive treatment for 1 year (~17 cycles).
  Interventions: Drug: pembrolizumab; Drug: Poly-ICLC

INTERVENTIONS:
Drug: pembrolizumab — 200mg pembrolizumab will be given intravenously on Day 1 of each 3-week cycle
  Other Names: MK-3475; Keytruda
Drug: Poly-ICLC — The maximum tolerated dose of Poly ICLC will be given twice weekly, in each 3-week cycle:
  Week 1, Days 1 and 4
  Week 2, Days 8 and 11
  Week 3, Days 15 and 18
  Other Names: polyinosinic-polycytidylic acid-polylysine-carboxymethylcellulose; Hiltonol

SUMMARY:
The main purpose of this study is to determine the dose of poly-ICLC that is safe and tolerable when it is combined with pembrolizumab in patients with colon cancer. This study will also evaluate how the combination of pembrolizumab and poly-ICLC activates the immune system in the patient's blood and inside the tumor; how it affects the size and number of tumor(s) in each patient; and how effective the combination is in patients with colon cancer that is unlikely to respond to pembrolizumab alone.

DETAILED DESCRIPTION:
Mismatch repair genes normally serve to fix the small glitches that occur when DNA is copied as cells divide. In 1993, researchers discovered that mutations in human mismatch repair genes play a key role in the development of certain forms of colorectal cancer; individuals who are deficient in these mismatch repair genes are at high risk for colorectal cancer. Accumulating evidence has shown that immunotherapy may be most effective against these cancers.

Programmed cell death protein 1, also known as PD-1, functions as an immune checkpoint, down-regulating the immune system by preventing the activation of T-cells, which in turn reduces autoimmunity and promotes self-tolerance. A new class of immunotherapy drugs that block PD-1, the PD-1 inhibitors, activate the immune system to attack tumors and are therefore used with varying success to treat some types of cancer.

Current clinical trials are showing that patients whose tumors are mismatch repair deficient are more likely to respond to immune-boosting anti-PD-1 drugs-such as pembrolizumab-than those with tumors proficient in mismatch repair. The idea is that the greater the number of DNA glitches in a tumor cell, the more abnormal proteins it will produce-and the more abnormal proteins that are generated, the greater the odds that the body's immune cells will regard the tumor cells as "foreign" and target them for destruction. Thus far, PD-1 inhibitors have shown great promise for mismatch repair deficient cancer patients, but not for mismatch repair proficient (MRP) cancer patients.

In this clinical trial, the investigators hypothesize that treating MRP colon cancer patients with immunostimulating agent poly-ICLC will generate an inflammatory response, increasing epitope recognition and development of tumor reactive T-cells at the tumor site. However, interferon alpha and gamma produced by the poly-ICLC will increase PD-L1 expression and limit new T-cell development. Thus, PD1 blockade will increase the effectiveness of treatment with pembrolizumab.

ELIGIBILITY:
Diagnosis/Condition for Entry into the Trial Phase 1 - Presence of histologically confirmed malignancy that has progressed following at least one therapy and able to be visualized on imaging. Measurable disease is not required. Patients with known targetable mutations must have progressive disease on the appropriated targeted drug therapy.

Phase 2 - Presence of MRP colon cancer that has progressed following at least two lines of therapy. Ten patients will be included who have disease that can be biopsied pre- and post-therapy.

Inclusion Criteria:

* Be willing and able to provide written informed consent for the trial
* Have measurable disease based on RECIST 1.1 (Phase 2)
* Be willing to provide tissue from a newly obtained core or excisional biopsy of a tumor lesion
* Have a performance status of 0 or 1 on the ECOG Performance Scale
* Have adequate organ function, according to screening labs performed within 10 days of treatment initiation
* Subjects of childbearing potential must be willing to use an adequate method of contraception for the course of the study through 120 days after the last dose of study medication

Exclusion Criteria:

* Currently participating/previously participated in a therapeutic study and received study therapy or used an investigational device within 4 weeks of the first dose of treatment
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment
* Has a known history of active TB (Bacillus Tuberculosis)
* Hypersensitivity to pembrolizumab or any of its excipients
* Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent
* Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies), active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis.
* Has active autoimmune disease that has required systemic treatment in the past 2 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2018-01-10 (Actual); Primary Completion 2022-07-29 (Actual); Study Completion 2022-07-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Asha Nayak, MD, Principal Investigator — Georgia Cancer Center at Augusta University; Sharad Ghamande, MD, Study Director — Georgia Cancer Center at Augusta University
Locations (1):
- Georgia Cancer Center at Augusta University, Augusta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase 1: Poly-ICLC: 1mg: Cohort 1: Participants were administrated 1mg Poly-ICLC intramuscularly (IM) twice weekly. Pembrolizumab was administrated 200 mg intravenously (IV) every 3 weeks (q3W)
- Phase 1: Poly-ICLC 2mg: Cohort 2: Participants were administrated 2mg Poly-ICLC intramuscularly (IM) twice weekly. Pembrolizumab was administrated 200 mg intravenously (IV) every 3 weeks (q3W)
- Phase 2: Poly-ICLC: 2mg: Cohort 3: Participants were administrated 2mg Poly-ICLC intramuscularly (IM) twice weekly. Pembrolizumab was administrated 200 mg intravenously (IV) every 3 weeks (q3W)
Period: Overall Study
Arm/Group | Phase 1: Poly-ICLC: 1mg | Phase 1: Poly-ICLC 2mg | Phase 2: Poly-ICLC: 2mg
Started | 8 | 10 | 24
Completed | 0 | 0 | 0
Not Completed | 8 | 10 | 24

BASELINE CHARACTERISTICS:
Groups:
- Phase 1: Poly-ICLC: 2mg: Cohort 2: Participants were administrated 2mg Poly-ICLC intramuscularly (IM) twice weekly. Pembrolizumab was administrated 200 mg intravenously (IV) every 3 weeks (q3W)
- Total: Total of all reporting groups
Arm/Group | Phase 1: Poly-ICLC: 1mg | Phase 1: Poly-ICLC: 2mg | Phase 2: Poly-ICLC: 2mg | Total
Number analyzed (Participants) | 8 | 10 | 24 | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 7 | 11 | 24
  >=65 years | 2 | 3 | 13 | 18
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 15 | 26
  Male | 2 | 5 | 9 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 5 | 2 | 10 | 17
  White | 3 | 7 | 14 | 24
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Phase 1: Determine the Maximum Tolerated Dose of Poly-ICLC That Can be Combined With Pembrolizumab
Description: A minimum of 3 participants will be treated at dose level 1 (1mg).
  * If 0 out of 3 participants experience dose limiting toxicities (DLT), then dose escalation will proceed to dose level 2 (2mg).
  * If 1 out of 3 participants experience DLT, a cohort of additional 3 participants will be assigned to the same dose level (1mg).
  * If 2 or more participants of 3 (or 6) experience DLT at dose level 1, then enrollment of participants will be stopped.
Time Frame: 12 months
Population: The safety population for this trial includes all participants who received at least one dose of the investigational product and excludes any participants who were screen fails.
Measure: Number; unit: mg
Groups:
- Phase 1: Poly-ICLC: 1 and 2 mg: Cohort 1: Participants were administrated 1mg Poly-ICLC intramuscularly (IM) twice weekly. Pembrolizumab was administrated 200 mg intravenously (IV) every 3 weeks (q3W)
  Cohort 2: Participants were administrated 2mg Poly-ICLC intramuscularly (IM) twice weekly. Pembrolizumab was administrated 200 mg intravenously (IV) every 3 weeks (q3W)
Arm/Group | Phase 1: Poly-ICLC: 1 and 2 mg
Number analyzed (Participants) | 14
mg | 2

2. Primary Outcome: Phase 1 and 2: Determine the Response Rate of Metastatic MRP Colon Cancer (That Has Progressed Following Two Lines of Therapy in the Metastatic Setting) to the Combination of Pembrolizumab and Poly-ICLC
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: From baseline to disease progression (Expected 12-24 months)
Population: The analysis population is the number of patients who received treatment. The outcome measure population below is determined by the number of patients within each dataset (each cohort) with complete response (CR) or partial response (PR) defined by RECIST criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1: Poly-ICLC: 1mg | Phase 1: Poly-ICLC 2mg | Phase 2: Poly-ICLC: 2mg
Number analyzed (Participants) | 7 | 7 | 17
Participants | 0 | 0 | 1

3. Primary Outcome: Determine the Overall Survival Rate for Recurrent Metastatic MRP Colon Cancer Response to the Combination of Pembrolizumab and Poly-ICLC
Description: The overall survival rate of response to the combination of pembrolizumab and poly-ICLC administered at the Recommended Phase 2 Dose (RP2D) will be estimated along with the correspondent 95% confidence interval.
Time Frame: From baseline to disease progression (up to 24 months)
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1: Poly-ICLC: 1mg | Phase 1: Poly-ICLC: 2mg | Phase 2: Poly-ICLC: 2mg
Number analyzed (Participants) | 8 | 10 | 24
Participants | 0 | 0 | 0

4. Secondary Outcome: Determine the Adverse Event Profile and Dose Limiting Toxicities of the Combination of Pembrolizumab and Poly-ICLC
Description: The adverse event profile will be presented by dose level of the combination treatment for the phase I portion
Time Frame: 12 months
Population: The percentage of participants that experienced severe adverse events.
Measure: Number; unit: percentage of participants
Arm/Group | Phase 1: Poly-ICLC: 1mg | Phase 1: Poly-ICLC 2mg | Phase 2: Poly-ICLC: 2mg
Number analyzed (Participants) | 8 | 10 | 24
percentage of participants | 87.5 | 70 | 70.83

5. Secondary Outcome: Determine the 20-week Progression Free Survival Rate of Recurrent Metastatic MRP Colon Cancer to the Combination of Pembrolizumab and Poly-ICLC
Description: The 20-week progression free survival rate for the combination of pembrolizumab and poly-ICLC administered at the Recommended Phase 2 Dose (RP2D) will be estimated along with the correspondent 95% confidence interval.
Time Frame: 20 weeks
Population: Progression is defined using Response Evaluation Criteria in Solid Tumors (RECIST v1.1) as any tumor enlargement greater than 20% and 5mm from baseline. The number of patients analyzed were the patients who received treatment. The outcome measure describes the count of patients who did not progress.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1: Poly-ICLC: 1mg | Phase 1: Poly-ICLC 2mg | Phase 2: Poly-ICLC: 2mg
Number analyzed (Participants) | 7 | 7 | 17
Participants | 0 | 0 | 0

6. Secondary Outcome: Determine the Duration of Response of Recurrent Metastatic MRP Colon Cancer to the Combination of Pembrolizumab and Poly-ICLC
Description: The duration of response to the combination of pembrolizumab and poly-ICLC administered at the Recommended Phase 2 Dose (RP2D) will be estimated along with the correspondent 95% confidence interval.
Time Frame: From baseline to disease progression (up to 24 months)
Population: Only one participant on this trial responded to the study treatment, so the 95% confidence interval could not be calculated.
Measure: Number; unit: weeks
Arm/Group | Phase 1: Poly-ICLC: 1mg | Phase 1: Poly-ICLC 2mg | Phase 2: Poly-ICLC: 2mg
Number analyzed (Participants) | 0 | 0 | 1
weeks |  |  | 36

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | Phase 1: Poly-ICLC: 1mg | Phase 1: Poly-ICLC: 2mg | Phase 2: Poly-ICLC: 2mg
All-Cause Mortality (participants affected / at risk) | 8/8 | 10/10 | 23/24
Serious Adverse Events (participants affected / at risk) | 7/8 | 7/10 | 17/24
Other Adverse Events (participants affected / at risk) | 0/8 | 0/10 | 0/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1: Poly-ICLC: 1mg (N=8) | Phase 1: Poly-ICLC: 2mg (N=10) | Phase 2: Poly-ICLC: 2mg (N=24)
Abdominal Distention (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 2 (2)
Small Bowel Obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1)
Death (General disorders) | 1 (1) | 1 (1) | 2 (2)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Intracranial Hemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Acute Kidney Injury (Renal and urinary disorders) | 1 (1) | 1 (1) | 1 (1)
Nausea/Vomitting (Gastrointestinal disorders) | 0 (0) | 1 (2) | 2 (2)
Thrombolytic Event (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperuricemia (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Tumor Lysis Syndrome (General disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Fever (General disorders) | 1 (1) | 0 (0) | 1 (1)
Malaise (General disorders) | 1 (1) | 0 (0) | 2 (2)
Fatigue (General disorders) | 1 (1) | 1 (1) | 0 (0)
Pulmonary Edema (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoglycemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Acute Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Hyponatrenia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Dehydration (General disorders) | 0 (0) | 1 (1) | 1 (1)
Blood Biliruben Increased (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2)
Hydrocephalis (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Abdominal Pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Kidney Infection (General disorders) | 0 (0) | 0 (0) | 1 (1)
Ascites (General disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2022-11-15): https://cdn.clinicaltrials.gov/large-docs/52/NCT02834052/Prot_SAP_ICF_001.pdf